CLINICAL TRIAL: NCT06910657
Title: A First-in-human, Phase I, Multi-center, Open-label, Dose-escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Preliminary Evidence of Antitumor Activity of IDOV-Immune in Adult Participants With Advanced Solid Tumors
Brief Title: IDOV-Immune for Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: ViroMissile, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VM-002-101
Record Dates: First submitted 2025-03-21; First posted 2025-04-04 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Colorectal Cancer; Pancreatic Cancer; Melanoma; Ovarian Cancer; Gastric Cancer; Esophageal Cancer; Hepatocellular Carcinoma; Renal Cell Carcinoma; Breast Cancer; Sarcoma; Bladder Cancer; Lung Cancer; Prostate Cancer; Cervical Cancers; Head and Neck Cancers; Adrenal Gland Tumors
Keywords: Oncolytic Virus Therapy; Advanced Solid Tumors; Metastatic Cancer; Refractory Cancer; Immunotherapy; Vaccinia Virus
MeSH Terms: conditions — Colorectal Neoplasms; Pancreatic Neoplasms; Melanoma; Ovarian Neoplasms; Stomach Neoplasms; Esophageal Neoplasms; Carcinoma, Hepatocellular; Carcinoma, Renal Cell; Breast Neoplasms; Sarcoma; Urinary Bladder Neoplasms; Lung Neoplasms; Prostatic Neoplasms; Uterine Cervical Neoplasms; Head and Neck Neoplasms; Adrenal Gland Neoplasms; Neoplasm Metastasis; Neoplasms; Vaccinia

STUDY DESIGN:
Intervention Model Description: This is a Phase I, open-label, single-group, dose-escalation study evaluating IDOV-Immune, an investigational oncolytic vaccinia virus, in adults with advanced solid tumors. Participants will receive a single intravenous (IV) infusion, with dose levels adjusted based on safety data using a Bayesian Optimal Interval (BOIN) design. The primary goal is to assess safety, tolerability, and determine the recommended Phase 2 dose (RP2D).
  Dose-limiting toxicities (DLTs) will be monitored for 28 days after dosing. Following dose escalation, expansion cohorts may be opened at selected doses to further evaluate safety and preliminary antitumor activity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- IDOV-Immune Dose Escalation Arm (Experimental): Participants in this arm will receive a single intravenous (IV) infusion of IDOV-Immune, an investigational oncolytic vaccinia virus, on Day 1 of a 28-day treatment cycle. The study will follow a dose-escalation design, with each successive cohort receiving an increased dose based on safety data and observed dose-limiting toxicities (DLTs). Following dose escalation, expansion cohorts may be enrolled at selected dose levels to further assess safety and preliminary antitumor activity.
  Interventions: Biological: IDOV-Immune (oncolytic vaccinia virus)

INTERVENTIONS:
Biological: IDOV-Immune (oncolytic vaccinia virus) — IDOV-Immune is a genetically engineered oncolytic vaccinia virus designed to selectively infect and destroy tumor cells while stimulating the immune system. This study investigates IDOV-Immune as a single intravenous infusion in a first-in-human, Phase 1, dose-escalation trial in participants with advanced solid tumors. The dose will escalate based on safety data, with a goal of identifying the recommended Phase 2 dose (RP2D).

SUMMARY:
This is a Phase I clinical trial evaluating an investigational treatment called IDOV-Immune, a type of oncolytic virus therapy, for adults with advanced solid tumors that have not responded to standard treatments. Oncolytic viruses are designed to infect and destroy cancer cells and have the potential to stimulate the immune system to fight the tumor.

The purpose of this study is to determine the safety of IDOV-Immune, how well it is tolerated, and to identify the highest dose that can be safely given. Researchers will also study how the drug behaves in the body, how the immune system responds to it, and whether it shows any signs of shrinking tumors.

Participants will receive a single intravenous (IV) infusion of IDOV-Immune and will be closely monitored for side effects and any changes in their cancer.

This study is being conducted at multiple sites in the United States and Australia.

DETAILED DESCRIPTION:
This is a first-in-human (FIH), Phase I, open-label, multi-center clinical trial designed to evaluate IDOV-Immune, an investigational oncolytic vaccinia virus-based immunotherapy, in adult participants with advanced solid tumors who have exhausted standard treatment options.

IDOV-Immune is a genetically engineered vaccinia virus designed to selectively infect and destroy tumor cells while enhancing immune responses through the expression of immune-stimulating molecules. It has been further modified to improve tumor selectivity and minimize the risk of harming healthy cells.

Study Design:

The trial will follow a dose-escalation design to determine the maximum tolerated dose (MTD), the recommended Phase 2 dose (RP2D), and the overall safety and tolerability profile of IDOV-Immune. A Bayesian Optimal Interval (BOIN) design will guide dose-escalation decisions, based on observed dose-limiting toxicities (DLTs) during a 28-day observation period after the initial dose. The study will also assess preliminary signs of antitumor activity at each dose level.

IDOV-Immune will be administered as a single intravenous (IV) infusion on Day 1 of a 28-day treatment cycle. Participants will undergo frequent safety assessments, including physical exams, laboratory tests, imaging studies, and immune response monitoring. Pharmacokinetics (how the virus behaves in the body), pharmacodynamics (how the virus impacts immune and tumor-related biomarkers), and immunogenicity (the body's immune response to the virus) will also be evaluated.

Planned Enrollment and Cohorts:

The study is expected to enroll up to approximately 42 participants in the dose-escalation phase. If appropriate, additional participants may be enrolled in backfill cohorts at selected dose levels to further assess the safety, biomarkers , and preliminary efficacy in specific populations. Across all study parts, total enrollment could reach approximately 78 participants.

Study Objectives:

The primary objective is to assess the safety and tolerability of IDOV-Immune and to determine the RP2D for future studies. Secondary objectives include evaluating how the investigational product moves through and affects the body (pharmacokinetics and pharmacodynamics), as well as initial signs of tumor response, including objective response rate (ORR), disease control rate (DCR), and progression-free survival (PFS).

Rationale:

There remains a significant unmet need for effective therapies for patients with advanced solid tumors who have progressed on or are intolerant to standard treatments. Oncolytic viruses have the potential for destroying cancer cells and activating anti-tumor immune responses. IDOV-Immune's multi-pronged design - combining direct oncolysis, immune recruitment, and immune system activation - aims to maximize therapeutic potential while maintaining an acceptable safety profile.

Study Locations:

The study will be conducted at multiple clinical sites in the United States and Australia with expertise in early-phase oncology trials and oncolytic virus therapies.

ELIGIBILITY:
Key Inclusion Criteria:

* Age ≥ 18 years.
* Histologically or cytologically confirmed advanced solid tumors that have progressed despite standard therapy, or for which no standard therapy exists.
* ECOG performance status ≤ 1.
* Measurable disease per RECIST v1.1.
* Adequate organ and bone marrow function.
* At least 28 days since major surgery, prior immunotherapy, or radiotherapy (with exceptions for minor procedures).
* Negative pregnancy test for women of childbearing potential.
* Agreement to use effective contraception during treatment and for 3 months after.
* Ability to provide informed consent and comply with study requirements.

Key Exclusion Criteria:

* Prior treatment with an oncolytic virus.
* Active or recent vaccinia virus infection or smallpox/monkeypox vaccination within 10 years.
* Active uncontrolled infection requiring systemic treatment.
* History of hepatitis B, hepatitis C, or HIV (unless meeting protocol-specific criteria).
* Unresolved ≥ Grade 2 toxicities from prior therapies (except hair loss or stable chronic conditions).
* Active or symptomatic autoimmune disease requiring systemic therapy.
* Active or untreated CNS metastases (unless stable per protocol).
* Significant cardiac disease (e.g., NYHA Class III/IV heart failure).
* Interstitial lung disease or prior pneumonitis requiring steroids.
* Conditions requiring chronic immunosuppressive therapy.
* Severe skin disorders or history of pancreatitis.
* Bleeding disorders or history of recent serious thromboembolic events.
* Any medical or psychiatric condition that could interfere with study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose-Limiting Toxicities (DLTs) | First 28 days after treatment (Cycle 1)
  Number of participants experiencing dose-limiting toxicities during the first 28 days after IDOV-Immune infusion, assessed using NCI CTCAE v5.0.
Number of Participants With Treatment-Emergent Adverse Events (TEAEs) | Up to 90 days post-treatment
  Count of participants who experience treatment-emergent adverse events after receiving IDOV-Immune.
Determination of Maximum Tolerated Dose (MTD) | Through completion of dose-escalation phase (~24 months)
  Identification of the highest dose level at which ≤ 30% of participants experience DLTs.
Determination of Recommended Phase 2 Dose (RP2D) | Through completion of dose-escalation and evaluation of all safety, PK/PD, and clinical activity data (~24 months)
  Dose selected based on totality of safety, PK, PD, and efficacy data.

SECONDARY OUTCOMES:
Peak Whole Blood Viral Genome Copy Number | Up to 28 days post-infusion
  Measurement of the highest detected viral genome copy number in whole blood after administration of IDOV-Immune.
Peak Serum Cytokine (IL-12 and CXCL9) Concentration | Up to 28 days post-infusion
  Measurement of the highest detected IL-12 and CXCL9 levels in serum after administration of IDOV-Immune.
Serum Cytokine (IFN-β, IFN-γ, IL-1β, IL-6, IL-10, TNF-α, and TGF-β1) Concentration | Up to 28 days post-infusion
  Measurement of serum cytokine levels as a pharmacodynamic marker following IDOV-Immune administration.
Objective Response Rate (ORR) | Up to 12 months
  Percentage of participants with a best overall response of complete response (CR) or partial response (PR), assessed per RECIST v1.1.
Duration of Response (DOR) | Up to 12 months
  Time from first documented objective response (CR or PR) to progression or death.
Disease Control Rate (DCR) | Up to 12 months
  Proportion of participants achieving CR, PR, or stable disease (SD) lasting at least 8 weeks.
Progression-Free Survival (PFS) | Up to 12 months
  Time from first dose to documented disease progression or death from any cause.
Overall Survival (OS) | Up to 12 months
  Time from first dose to death from any cause.
Incidence of Neutralizing Antibody Response | Up to 90 days post-treatment
  Number of participants who develop detectable anti-vaccinia neutralizing antibodies after IDOV-Immune infusion.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (3):
  - Washington University School of Medicine, St Louis, Missouri
  - MD Anderson Cancer Center, Houston, Texas
  - South Texas Accelerated Research Therapeutics, San Antonio, Texas
- Australia (3):
  - Royal North Shore Hospital, Saint Leonards, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - The Alfred Hospital, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: Undecided